CLINICAL TRIAL: NCT00759590
Title: Comparisons of Two Methods to Estimate the Lung Recruitment
Brief Title: Comparison of Two Methods to Estimate the Lung Recruitment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 584
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ALI/ARDS patients
  Interventions: Procedure: CT scan and Pressure volume curve

INTERVENTIONS:
Procedure: CT scan and Pressure volume curve — CT scan

SUMMARY:
In this study the investigators aim to compare two common methods to estimate the lung recruitment in ALI/ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* ALI/ARDS

Exclusion Criteria:

* Barotrauma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALI/ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Study Chair — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy

REFERENCES:
- [Derived] Chiumello D, Marino A, Brioni M, Cigada I, Menga F, Colombo A, Crimella F, Algieri I, Cressoni M, Carlesso E, Gattinoni L. Lung Recruitment Assessed by Respiratory Mechanics and Computed Tomography in Patients with Acute Respiratory Distress Syndrome. What Is the Relationship? Am J Respir Crit Care Med. 2016 Jun 1;193(11):1254-63. doi: 10.1164/rccm.201507-1413OC. PMID 26699672